CLINICAL TRIAL: NCT00125723
Title: A Multicenter, Open-label, Phase 4 Study of Pegfilgrastim Administered in the First and Subsequent Cycles of Myelosuppressive Chemotherapy
Brief Title: FIRST - Study of Pegfilgrastim Administered in the First and Subsequent Cycles of Myelosuppressive Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030218
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Neutropenia
Keywords: Phase 4 Clinical Trial; Chemotherapy; Neulasta®; Oncology; Malignancy
MeSH Terms: conditions — Neutropenia; Neoplasms

ARMS (2):
- No Intervention (No Intervention)
  Interventions: Other: PI Discretion
- Intervention (Other): PI Discretion
  Interventions: Other: PI Discretion

INTERVENTIONS:
Other: PI Discretion — PI Discretion

SUMMARY:
The purpose of the study is to assess the impact of first and subsequent cycle pegfilgrastim on neutropenia events (such as hospitalizations, dose reductions and delays) in patients receiving myelosuppressive chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Pathologically confirmed diagnosis of the following malignancies: breast, non-Hodgkin's lymphoma (NHL), Hodgkin's disease, ovarian, colorectal, lung or other - Planned administration of a new myelosuppressive every 14 (q14), q21, or q28 day chemotherapy - Written informed consent for participation in the study before any study-specific procedures are performed, including screening and registration Exclusion Criteria: - Planned concomitant therapeutic radiation - Diagnosis of acute or chronic leukemia or myelodysplastic syndrome - Prior stem-cell transplantation (includes bone-marrow transplantation) - Medical diagnosis of chronic neutropenia of any cause not related to cancer - Current cytotoxic, biologic, or immunologic therapy for unrelated conditions - Subject has active infection requiring treatment - Known HIV-positive subjects - Subject of child-bearing potential is evidently pregnant (e.g., positive HCG test) or is breast feeding - Subject of child-bearing potential is not using adequate contraceptive precautions - Known sensitivity to E. coli derived drug products (e.g., filgrastim, HUMULIN® insulin, L-asparaginase, HUMATROPE® growth hormone, INTRON A®) - Any psychiatric, addictive or other kind of disorder which compromises the ability of the subject to give written informed consent and/or to comply with study protocol procedures - Subject is currently enrolled in, or has not yet completed at least 30 days since ending another device or drug trial(s) or is receiving, or plans to receive, other investigational agent(s) not approved by the Food and Drug Administration (FDA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2252 (Actual)
Dates: Start 2004-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
dose delays and dose reductions and neutropenic events | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Noga SJ, Choksi JK, Ding B, Dreiling L, Ozer H. Low incidence of neutropenic events in patients with lymphoma receiving first-cycle pegfilgrastim with chemotherapy: results from a prospective community-based study. Clin Lymphoma Myeloma. 2007 May;7(6):413-20. doi: 10.3816/CLM.2007.n.020. PMID 17621407
- [Result] Ozer H, Mirtsching B, Rader M, Luedke S, Noga SJ, Ding B, Dreiling L. Neutropenic events in community practices reduced by first and subsequent cycle pegfilgrastim use. Oncologist. 2007 Apr;12(4):484-94. doi: 10.1634/theoncologist.12-4-484. PMID 17470691
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20030218.pdf